CLINICAL TRIAL: NCT06185530
Title: Stress Echocardiography With Carotid Ultrasound vs Routine CT Coronary Angiography in Suspected Chronic Coronary Syndrome for the Detection of Obstructive Coronary Disease and Prevention of Adverse Outcomes.
Brief Title: SECURE Trial: Stress Echocardiography With Carotid Ultrasound vs Routine CT Coronary Angiography in Chronic Coronary Syndrome for Endpoints
Acronym: SECURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRC/2023/001
Record Dates: First submitted 2023-05-31; First posted 2023-12-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Chronic Coronary Syndrome; Coronary Disease; Coronary Artery Disease
Keywords: CTCA; Stress Echocardiography; Carotid Ultrasound
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants undergo the cardiac tests: stress echocardiography with carotid ultrasound (Experimental)
  Interventions: Diagnostic Test: Detection of obstructive coronary disease
- Participants undergo the cardiac test: CT coronary angiography (Active Comparator)
  Interventions: Diagnostic Test: Detection of obstructive coronary disease

INTERVENTIONS:
Diagnostic Test: Detection of obstructive coronary disease — Detection of obstructive coronary disease

SUMMARY:
Diseases of the heart and circulation are known as cardiovascular diseases, and they cause over 160,000 deaths each year.

Coronary heart disease (CHD) is the most common cardiovascular disease. This is due to a build-up of fatty material, known as atherosclerosis, in the blood vessels supplying blood to the heart muscle. This can cause chest pain or if blocked, can cause a heart attack.

Two of the main non-invasive tests to look for coronary heart disease are Computed Tomography Coronary Angiography (CTCA) and Stress Echocardiography (Ultrasound scan).

CTCA shows the arteries and allows small amounts of disease to be seen that may not yet be causing any symptoms. However, if there's lots of disease and calcification, it becomes difficult to tell how severe it is, which means several tests may be needed. Stress Echocardiography shows if enough blood is reaching the heart muscle, so can show if there is severe disease that needs treatment. However, it can't see the arteries so doesn't showt small disease that may benefit from tablet treatment. There is not yet an effective non-invasive combined test that can give all this information in one go.

Studies have shown that if there's atherosclerosis in another artery, a person is very likely to have coronary atherosclerosis as well. Carotid atherosclerosis, in the neck arteries, can be seen with ultrasound similar to stress echocardiography. So, by combining these two tests the investigators want to see if it is possible to see severe as well as small areas of disease in one test, to provide better treatment.

The study will enrol 2,000 participants, who need investigation for CHD, equally randomised to CTCA or stress echocardiography with carotid ultrasound. We will follow these participants for 5 years and observe for any adverse outcomes and ask them to complete a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Patients referred to RACPC and judged by the reviewer to require a further imaging investigation, either SE or CTCA, to evaluate a suspected diagnosis of CAD
3. AND

   1. Have a PTP score ≥ 5%, as calculated using ESC guidelines OR
   2. Have clinical history in keeping with 'typical' angina symptoms, as judged by the investigator, in patients with a PTP score <5% - With 'typical' symptoms, as per ESC guidelines, being all three of the following

   i) Constricting symptoms in the front of the chest or in the neck, jaw, shoulder or arm ii) Precipitated by physical exertion iii) Relieved by rest or nitrates within 5 minutes
4. Able to give informed consent to participate in the study and its follow up

Exclusion Criteria:

1. Patients with diagnosed ACS that require urgent or emergency treatment or hospitalisation for inpatient investigations.
2. Known history of obstructive CAD (Previous MI, PCI or CABG) or previous invasive angiography with evidence of ≥ 50% stenosis in any epicardial vessel.
3. Patients who have undergone invasive or non-invasive, functional or anatomical (Including CAC score) testing for detection of CAD within the previous 1 year of clinical assessment.
4. Documented allergy to iodinated contrast or documented allergy to both ultrasound contrasts used at LNWH Trust; Luminity® (Perflutren) and SonoVue® (Sulphur Hexafluoride) or the constitutes
5. Contraindications to undergoing CTCA, including but not limited to;

   * eGFR < 40 ml/min
   * Contraindications to beta-blockers including but not limited to, documented allergy or significant airways disease in the judgement of the investigator.
   * Exceeding CT scanner weight tolerance
6. Contraindications to undergoing SE, including but not limited to;

   * Known cardiomyopathic process (Hypertrophic cardiomyopathy (HCM)) with resting gradient > 50mmHg or severe valvular lesion
   * Severe uncontrolled hypertension (≥180/100mmHg)
7. Known pregnancy
8. Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of obstructive CAD and prevalence of MACE in enrolled participants | Within 3 months of randomisation confirmed by documentation in medical record

SECONDARY OUTCOMES:
Assessment of resource utilisation between study arms (subsequent downstream testing, cardiac related hospital visits, costs and incremental cost effectiveness) | Time to first event, up to 18 months post randomisation, confirmed by medical record documentation
Assessment of overall ionising radiation exposure (dose) between study arms | Within 3 months of randomisation, confirmed by documentation in investigation report
Major complications from cardiovascular procedures or cardiovascular diagnostic testing | Up to18 months from randomisation to time of first documented outcome in medical records
  (a. Haemodynamically unstable new arrhythmia requiring emergency respiratory and/or circulatory support b. Anaphylaxis defined as a new severe reaction requiring emergency respiratory and/or circulatory support to administration of medication, including but not limited to; iodinated contrast, ultrasound contrast, dobutamine or atropine.
  c. Major bleeding requiring a transfusion of ≥ 1 unit of packed red blood cells and/or further interventional procedures related to bleeding management.
  d. Acute severe renal failure requiring ≥ 1 cycle of renal replacement therapy. e. Stroke defined as sudden onset focal neurological deficit with cerebral imaging confirming new stroke)
Analysis of patient derived chest pain related quality of life (EQ-5D) | at 6-months and 12-months after randomisation on telephonecall questionnaire completion with patient
Change in prescription of preventative therapies (including statin and anti-platelet agents or dose increase of current statin therapy > 50%) | Up to 18 months from randomisation to time of first documented outcome in medical records
The proportion of patients undergoing invasive coronary angiography and revascularisation, of the target lesion, either through PCI or CABG, at follow up. | Time (in days) from the initial investigation until revascularisation confirmed by medical record documentation

CONTACTS AND LOCATIONS:
Overall Officials: Prof Roxy Senior, Principal Investigator — LNWH Trust
Locations (1):
- London North West University Healthcare NHS Trust, Harrow, Middx, United Kingdom

IPD SHARING:
Plan to Share IPD: No